CLINICAL TRIAL: NCT00341627
Title: Genetic Aspects of Chordoma: A Collaboration With SEER Registries to Identify Chordoma Families
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999005; OH99-C-N005
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chordoma
Keywords: Bone Tumor; Familial Chordoma; Gene Mapping; Genetics; Sporadic Chordoma
MeSH Terms: conditions — Chordoma; Bone Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Population-based sampling of individuals affected with Chordoma

SUMMARY:
Chordoma is an uncommon (400 case/year in the U.S.) and potentially fatal bone tumor derived from remnants of embryonic notochord. It occurs primarily in the axial skeleton and has a mean age at diagnosis of 55 years, with a range from early childhood to over 70 years. This tumor usually presents at an advanced stage and the associated mortality is high due to local destruction and distant metastases. Chordoma is rare in African-Americans and is typically sporadic; there are few reports of these tumors arising congenitally or within members of the same family.

Recently, we have identified and studied one large family in which 10 relatives in three generations have chordoma; the inheritance pattern suggests transmission of a mutation in an autosomal dominant gene. Using information from this family, we have tentatively napped this gene to the long arm of chromosome 7. To confirm this finding, and to fine map and clone the gene, we need to study additional chordoma families. In an effort to identify such families, we have developed collaborations with four SEER registries covering the populations of Detroit, Los Angeles, Iowa, and New Mexico. Each registry will identify all chordoma cases diagnosed since 1988 and invite them (or the next of kin of deceased cases) to participate in our study. Through 1997, the registries have identified a total of 140 chordoma cases, 96 of whom are living. The registries will invite these patients (or their next of kin) to participate in the study. The study components include completion of a self-administered personal and family medical history questionnaire, retrieval of medical records and pathology reports pertaining to chordoma, and collection of paraffin-embedded chordoma tissue and buccal mucosal cells for genetic studies. NCI will carry out all the data collection activities for the study subjects identified through the Detroit registry. NCI will also conduct the buccal cell collection component of the study for all patients identified by the other three registries. These three registries will carry out all other study activities on these patients/next of kin and will send the data and slides prepared from the paraffin blocks to NCI. NCI will analyze the questionnaire data to determine if any unusual patterns of cancers other than chordoma or other medical conditions appear to cluster in families of the chordoma patients. Selected members of any families with two or more relatives with chordoma will be invited to participate in a separate clinical and molecular study conducted at NIH to try to identify the chordoma gene. DNA from the buccal cells and tumor blocks from all other patients with "sporadic" chordoma identified through the registries (likely to comprise most patients) will not be studied until we or others have identified such a gene.

DETAILED DESCRIPTION:
Chordoma is an uncommon (400 case/year in the U.S.) and potentially fatal bone tumor derived from remnants of embryonic notochord. It occurs primarily in the axial skeleton and has a mean age at diagnosis of 55 years, with a range from early childhood to over 70 years. This tumor usually presents at an advanced stage and the associated mortality is high due to local destruction and distant metastases. Chordoma is rare in African-Americans and is typically sporadic; there are few reports of these tumors arising congenitally or within members of the same family.

In 1996, we have identified and studied one large family in which 8 relatives in three generations have chordoma; the inheritance pattern suggests transmission of a mutation in an autosomal dominant gene. Using information from this family, we tentatively mapped this gene to the long arm of chromosome 7. To confirm this finding, and to fine map and clone the gene, we needed to study additional chordoma families.

In an effort to identify such families, we have developed collaborations with four SEER registries covering the populations of Detroit, Los Angeles, Iowa, and New Mexico. Each registry will identify all chordoma cases diagnosed since 1988 and invite them (or the next of kin of deceased cases) to participate in our study. Through 1997, the registries have identified a total of 140 chordoma cases, 96 of whom are living. The registries will invite these patients (or their next of kin) to participate in the study. The study components included completion of a self-administered personal and family medical history questionnaire, retrieval of medical records and pathology reports pertaining to chordoma, and collection of paraffin-embedded chordoma tissue and buccal mucosal cells for genetic studies. NCI carried out all the data collection activities for the study subjects identified through the Detroit registry. NCI also conducted the buccal cell collection component of the study for all patients identified by the other three registries. These three registries will carry out all other study activities on these patients/next of kin and sent the data and slides prepared from the paraffin blocks to NCI. NCI will analyze the questionnaire data to determine if any unusual patterns of cancers other than chordoma or other medical conditions appear to cluster in families of the chordoma patients. Selected members of any families with two or more relatives with chordoma will be invited to participate in a separate clinical and molecular study conducted at NIH to try to identify the chordoma gene. DNA from the buccal cells and tumor blocks from all other patients with 'sporadic' chordoma identified through the registries (likely to comprise most patients) will not be studied until we or others have identified such a gene.

ELIGIBILITY:
* INCLUSION CRITERIA:

All persons with chordoma reported to the four tumor registries from January 1988 to the end of the study period.

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population-based sampling of individuals affected with Chordoma
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 1999-02-01 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Identification of families containing multiple cases of Chordoma. | Ongoing
  To determine if any unusual patterns of cancers other than chordoma or other medical conditions appear to cluster in families of the chordoma patients with the ultimate, long-term goal fine-mappingthe gene(s) involved in chordoma.

CONTACTS AND LOCATIONS:
Overall Officials: Mary L McMaster, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - NCI, DCEG, Clinical Genetics Branch, Rockville, Maryland

REFERENCES:
- [Background] Yang X', Beerman M, Bergen AW, Parry DM, Sheridan E, Liebsch NJ, Kelley MJ, Chanock S, Goldstein AM. Corroboration of a familial chordoma locus on chromosome 7q and evidence of genetic heterogeneity using single nucleotide polymorphisms (SNPs). Int J Cancer. 2005 Sep 1;116(3):487-91. doi: 10.1002/ijc.21006. PMID 15818627
- [Background] Yang XR, Ng D, Alcorta DA, Liebsch NJ, Sheridan E, Li S, Goldstein AM, Parry DM, Kelley MJ. T (brachyury) gene duplication confers major susceptibility to familial chordoma. Nat Genet. 2009 Nov;41(11):1176-8. doi: 10.1038/ng.454. Epub 2009 Oct 4. PMID 19801981
- [Background] Kelley MJ, Shi J, Ballew B, Hyland PL, Li WQ, Rotunno M, Alcorta DA, Liebsch NJ, Mitchell J, Bass S, Roberson D, Boland J, Cullen M, He J, Burdette L, Yeager M, Chanock SJ, Parry DM, Goldstein AM, Yang XR. Characterization of T gene sequence variants and germline duplications in familial and sporadic chordoma. Hum Genet. 2014 Oct;133(10):1289-97. doi: 10.1007/s00439-014-1463-z. Epub 2014 Jul 4. PMID 24990759